CLINICAL TRIAL: NCT02347943
Title: OASIS Global Sinus Surgery Registry
Brief Title: Global Sinus Surgery Registry
Acronym: OASIS
Status: Terminated | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR005044
Record Dates: First submitted 2015-01-19; First posted 2015-01-28 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Chronic Rhinosinusitis; Recurrent Acute Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates long-term safety and effectiveness of primary sinus surgery in a real-world population of adults with chronic rhinosinusitis (CRS) or recurrent acute rhinosinusitis (RARS). This post-market study will evaluate sinus surgery performed using commercially available sinus instrumentation (e.g. sinus balloon catheters, powered microdebriders, manual instruments).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum adult age as required by local regulations
* The subject has a planned primary sinus surgery, which includes either traditional transnasal endoscopic sinus surgery (ESS), balloon sinus dilation (BSD) or a hybrid procedure
* Subjects diagnosed by ENT surgeon with chronic rhinosinusitis (CRS) or recurrent acute rhinosinusitis (RARS) per AAO-HNS or EPOS adult sinusitis clinical practice guidelines
* The subject has been informed of the nature of the registry and has consented to participate and authorized the collection and release of medical information by signing a consent form
* Subject is able to read and understand local language

Exclusion Criteria:

* Prior sinus surgery. Septoplasty, Nasal Polypectomy, Septorhinoplasty, Nasal Valve and Turbinate Reduction surgeries are not exclusions
* Planned surgery of any of the following : orbital decompression, skull base, neoplasm, lacrimal, UPPP, aesthetic surgery, Potts Puffy tumor, Draf III
* Planned external approaches (i.e. not trans-nasal)
* Planned off-label usage of balloon sinus dilation products.
* Balloon sinus dilation performed with a non-Acclarent balloon product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed by an ENT surgeon with chronic rhinosinusitis (CRS) or recurrent acute rhinosinusitis (RARS) undergoing a primary transnasal endoscopic sinus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Phoenix, Arizona
  - Los Angeles, California
  - Sacramento, California
  - San Francisco, California
  - Miami, Florida
  - Atlanta, Georgia
  - Evans, Georgia
  - Berwyn, Illinois
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - West Burlington, Iowa
  - Alexandria, Louisiana
  - Bethesda, Maryland
  - City of Saint Peters, Missouri
  - Helena, Montana
  - Henderson, Nevada
  - Albuquerque, New Mexico
  - Long Beach, New York
  - New York, New York
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - McKinney, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Sinus Dilation: Subjects who underwent a balloon sinus dilation procedure
- Endoscopic Sinus Surgery (ESS): Subjects who underwent a transnasal endoscopic sinus surgery
- Hybrid: Subjects who underwent a procedure with balloon sinus dilation and transnasal endoscopic sinus surgery.
Period: Overall Study
Arm/Group | Balloon Sinus Dilation | Endoscopic Sinus Surgery (ESS) | Hybrid
Started | 140 | 67 | 45
Completed | 0 | 0 | 0
Not Completed | 140 | 67 | 45
Not completed — Study was cancelled | 140 | 67 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balloon Sinus Dilation | Endoscopic Sinus Surgery (ESS) | Hybrid | Total
Number analyzed (Participants) | 140 | 67 | 45 | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (14.83) | 43.3 (14.42) | 43.8 (18.02) | 45.5 (15.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 39 | 29 | 145
  Male | 63 | 28 | 16 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 9 | 34
  Not Hispanic or Latino | 127 | 55 | 36 | 218
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 1 | 1 | 2 | 4
  Black or African American | 16 | 0 | 2 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 3 | 0 | 5 | 8
  White | 118 | 64 | 36 | 218

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Follow-Up Visits
Time Frame: 2 years
Population: Due to early cancellation of the study data for this endpoint were not collected.
Groups:
- Endoscopic Sinus Surgery: Subjects who underwent a transnasal endoscopic sinus surgery
Arm/Group | Balloon Sinus Dilation | Endoscopic Sinus Surgery | Hybrid
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Balloon Sinus Dilation (BSD): Subjects who underwent a balloon sinus dilation procedure
Arm/Group | Balloon Sinus Dilation (BSD) | Endoscopic Sinus Surgery (ESS) | Hybrid
Serious Adverse Events (participants affected / at risk) | 1/140 | 1/67 | 0/45
Other Adverse Events (participants affected / at risk) | 8/140 | 4/67 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (BSD) (N=140) | Endoscopic Sinus Surgery (ESS) (N=67) | Hybrid (N=45)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (BSD) (N=140) | Endoscopic Sinus Surgery (ESS) (N=67) | Hybrid (N=45)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dehiscence in the lamina papyracea (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the early cancellation of the study, study results reported are limited to subject enrollment, subject demographics, and Adverse Events (SAE and Non-serious).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No